CLINICAL TRIAL: NCT07234656
Title: Patient-partnered Research: a Key to Investigating Fear of Cancer Recurrence in Patients With Surgically Treated Kidney Cancer (PP-RECURK)
Brief Title: Patient-partnered Research in Investigating Fear of Cancer Recurrence in Kidney Cancer
Acronym: PP-RECURK
Status: Recruiting | Type: Observational
Sponsor: Brigitta Rasmussen Villumsen (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Brigitta Rasmussen Villumsen, Principal Investigator, Gødstrup Hospital
Organization: Gødstrup Hospital (Other)
Other Study IDs: 1-16-02-314-25
Record Dates: First submitted 2025-08-06; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Fear of Cancer Recurrence; Renal Cell Carcinoma (Kidney Cancer)
Keywords: Fear of Cancer Recurrence; Patient involvement in research; Kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Panel members: 6 patients with spouses/partners and 3 single patients. In total 15 subjects.
  Interventions: Other: Phase 1: Establishment of a patient-partner panel
- Pilot population: In total 90 subjects (patients with or without partners)
  Interventions: Other: Phase 2: Feasibility testing of FCR questions, mode of administration and timing for investigating Fear of Cancer Recurrence

INTERVENTIONS:
Other: Phase 1: Establishment of a patient-partner panel — Phase 1: Establishment of a patient-partner panel who in collaboration with researchers define Fear of Cancer Recurrence questions, mode of administration and timing for investigating Fear of Cancer Recurrence in phase 2 (pilot testing in a feasibility study).
  Groups: Panel members
Other: Phase 2: Feasibility testing of FCR questions, mode of administration and timing for investigating Fear of Cancer Recurrence — As the intervention for phase 2 is a product of the collaboration and discussions between panel members and researchers during phase 1, the intervention can not be described more detailed.
  Groups: Pilot population

SUMMARY:
The goal of this observational study is to gather real-world information about Fear of Cancer Recurrence (FCR) following surgery in patients with renal cell carcinoma (RCC) and their partners/spouses by 1) establishing a panel consisting of patients with or without partners/spouses to facilitate patient-partnered research. Furthermore, 2) Through discussions among panel members and researchers identification of the most pertinent topics related to FCR, as well as the optimal timing and methods for collecting that information in the follow-up care after surgery. Finally, to conduct a feasibility and pilot study to investigate the feasibility of the recommendations developed in 1) + 2) and assess FCR in patients with RCC following surgery and their partners/spouses.

In phase 1 participants (panel members) will be asked to collaborate with researchers in the development of recommendations for FCR questions, mode of administration and timing in the follow-up care after surgically treated kidney cancer.

In phase 2 participants (patients and partners) in follow-up care after surgically treated kidney cancer are asked to answer questions about FCR at specific timepoints defined by panel members and researchers in phase 1.

DETAILED DESCRIPTION:
Rationale Previously, Fear of Cancer Recurrence (FCR) has been investigated in patients with renal cell carcinoma (RCC) showing that FCR is the most common source of frustration, and the prevalence of FCR has been estimated to be 54% in patients with localized RCC.

Studies in families with cancer show that approximately 50% of family caregivers experience FCR.

Patient involvement in research is much requested, however, no study to date has involved patients and partners/spouses in the investigation of FCR in patients with kidney cancer and their family caregivers.

Therefore, in this study the investigators will ask patients with localized kidney cancer and their partners/spouses to contribute with their perspectives on what questions to ask in the follow-up care after surgery for kidney cancer to identify FCR. For this purpose, the validated 42-item Fear of Cancer Inventory (FCRI) will be used for inspiration. A caregiver version of the FCRI exists, but has not been translated to Danish and thus translation will be conducted in this study.

This study is expected to provide information to clinicians on how to comply with the European Association of Urology guideline that recommends psychological evaluation for all patients diagnosed with RCC and involvement of patients in adjuvant RCC treatment decisions. Furthermore, the investigators conduct this study to give patients with kidney cancer and partners/spouses a voice in the investigation of FCR in the clinical follow-up care after surgery. This provides an opportunity for a collaboration between patients, partners, patients associations and professional researchers to identify the most appropriate FCR questions, timing, and mode of administration to optimize patient adherence/compliance and treatment outcomes.

Method The project has two phases. Phase 1: Establishment of a patient/partner panel who in collaboration with researchers will use the 5-stage Design thinking model to develop recommendations for investigating FCR in patients and their partners/spouses in follow-up care after surgically treated kidney cancer.

The Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework described by Glasgow et al. will be applied for the process evaluation of recruitment and eligibility of panelists.

The level of meaningful patient/partner/spouse engagement in the project will be evaluated using the Patient Engagement in Research Scale (PEIRS-22).

Phase 2:

The recommendations produced in phase 1 will be tested in a pilot and feasibility study along with investigation of additional factors possibly affecting fear of cancer recurrence in patients and their partners/spouses. All evaluations will be done statistically.

Perspectives If the phase 2 pilot-study turns out successfully in defining FCR in patients with RCC and their partners/spouses, the researchers will seek to perform a national follow-up study, that can constitute a foundation for implementation of FCR as part of standard clinical practice, e.g. detecting when FCR reaches a level that needs interference such as psychological counselling etc.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

* Single patients diagnosed with Renal Cell Carcinoma (RCC) or patients with RCC being in an intimate relationship with a partner/spouse
* Partner/spouse to patients who fullfil the inclusion criteria
* Patients have undergone surgery due to localized RCC (T1-T2-T3 tumor)
* Time since surgery: 0-120 months
* Danish speaking patients and partners/spouses. Must be able to speak, write and read Danish
* Patients/partners/spouses able to and willing to attend online project meetings or in person at Gødstrup Hospital.

Phase 2:

* Single patients diagnosed with Renal Cell Carcinoma (RCC) or patients with RCC being in an intimate relationship with a partner/spouse
* Partner/spouse to patients who fullfill the inclusion criteria
* Patients who have undergone surgery due to localized RCC (T1-T2-T3 tumor)
* Danish speaking patients and partners/spouses. Must be able to speak, write and read Danish
* Able to receive digital communication from the hospital
* Informed consent must be signed before answering Fear of Cancer Recurrence questions

Exclusion Criteria:

Both phases, both patients and partners/spouses:

* Diagnosed with cognitive impairment
* Untreated psychiatric disorders due to non-compliance

Phase 2:

• Patients and partners/spouses who were panelists in phase 1

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and partners who fullfil the in- and exclusion criteria and are consulting urologists at Aalborg University Hospital, Aarhus University Hospital and Gødstrup Hospital, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Assessment of the recruitment to and composition the patient-partner panel | From inclusion to week 16 or date of last subject included whichever comes first.
  The RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework will be applied for the assessment of the recruitmentprocess, eligibility of panelists and their representativity.
Phase 1: Assessment of the degree of patient and partner/spouse involvement | From inclusion to week 26 or end of engagement whichever comes first.
  The Patient Engagement in Research Scale (PEIRS) will be applied to assess the degree of meaningful patient and family caregiver engagement in research from a patient and partner/spouse perspective.
  The 22-item Patient Engagement in Research Scale (PEIRS) score ranges from 0-88. Minimum value per item: 0 (Strongly Disagree), maximum value per item: 4 (Strongly Agree). Higher scores = better engagement in research.
  To make interpretation easier, many studies convert the raw total to a 0-100 score calculated by taking the total sum score, divided by 88 (22 items X 4 scores), and multiplying it by 100
Phase 2: To investigate whether the recommendations for timing, instructions, mode of administration and Fear of Cancer Recurrence questions stated in phase 1 are feasible in a clinical setting, | From inclusion to week 52.
  Patients' and partners/spouses' compliance to the investigation of Fear of Cancer Recurrence will be evaluated using descriptive statistics.
  Fulfillment of the feasibility criteria are met when 80% of the included subjects complete the pilot testing.
Phase 2: The prevalence of Fear of Cancer Recurrence in single patients with localized Renal Cell Carcinoma | From inclusion to week 52 or when the subject withdraws from the study whichever comes first.
  Descriptive statistics will be used to present the level of Fear of Cancer Recurrence. Data will be presented as median Fear of Cancer Recurrence score with 95% Confidence Interval.
Phase 2: The prevalence of Fear of Cancer Recurrence in patients with localized Renal Cell Carcinoma and living in a relationship with a partner/spouse. | From inclusion to week 52 or when the subject withdraws from the study whichever comes first.
  Descriptive statistics will be used to present the level of Fear of Cancer Recurrence. Data will be presented as median Fear of Cancer Recurrence score with 95% Confidence Interval.
Phase 2: The prevalence of Fear of Cancer Recurrence in partners/spouses to patients with localized Renal Cell Carcinoma. | From inclusion to week 52 or when the subject withdraws from the study whichever comes first.
  Descriptive statistics will be used to present the level of Fear of Cancer Recurrence. Data will be presented as median Fear of Cancer Recurrence score with 95% Confidence Interval.

SECONDARY OUTCOMES:
Phase 2: Associations between data on Fear of Cancer Recurrence and disease stage in single patients. | From inclusion to week 52.
  Logistic regression analysis will be conducted to investigate associations between Fear of Cancer Recurrence and disease stage: Leibovich disease risk groups (low, medium, and high) .
  The Fear of Cancer Recurrence Inventory will be used to measure Fear of Cancer Recurrence (FCR). Higher score means higher FCR. The score range from 0-168.
Phase 2: Associations between data on Fear of Cancer Recurrence and comorbidity burden in single patients. | From inclusion to the study to week 52 or when the subject withdraws consent whichever comes first.
  Logistic regression analysis will be conducted to investigate associations between Fear of Cancer Recurrence and Charlson Comorbidity Index score.
  The Fear of Cancer Inventory will be used to measure FCR. Higher score means higher FCR. The score ranges from 0-168.
Phase 2: Associations between data on Fear of Cancer Recurrence and sex in single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and age in single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and educational level in single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and disease stage in patients with a partner/spouse. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and comorbidity burden in patients with a partner/spouse. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations between Fear of Cancer Recurrence score and Charlson Comorbidity Index score.
Phase 2: Associations between data on Fear of Cancer Recurrence and sex in patients with a partner/spouse. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and age in patients with a partner/spouse. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and educational level in patients with partner/spouse. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and patients' disease stage in partners/spouses of non-single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations between data on Fear of Cancer Recurrence and patients' disease stage: Leibovich disease risk groups (low, medium, and high).
Phase 2: Associations between data on Fear of Cancer Recurrence and partners'/spouses' comorbidities in partners/spouses of non-single patients. | From inclusion to week 52.
  Logistic statistical analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and sex of partners/spouses among non-single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and age of partners/spouses among non-single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.
Phase 2: Associations between data on Fear of Cancer Recurrence and educational level in partners/spouses of non-single patients. | From inclusion to week 52.
  Logistic regression analyses will be conducted to investigate associations.

OTHER OUTCOMES:
Phase 2: Investigate the association between Fear of Cancer Recurrence within couples (patient and partner/spouse). | From inclusion to week 52.
  For the investigation of the association between Fear of Cancer Recurrence (FCR) within couples (patient and partner) ideally the Actor-Partner Interdependence Model (APIM) will be applied. Alternatively, a Multilevel Model (MLM) can be applied if couples are treated as clusters to account for the dependent FCR scores between partners/spouses.
  The Fear of Cancer Inventory will be used to determine FCR. Higher score represents higher level of FCR. The score ranges from 0-168.
Phase 2: Comparison between Fear of Cancer Regression in single patients and patients living in a relationship. | From inclusion to week 52.
  To compare the Fear of Cancer Recurrence score between single patients and patients in relationship, the Mann-Whitney U test will be applied.
  The Fear of Cancer Inventory will be used to to determine FCR. Higher score represents higher level of FCR. The score ranges from 0-168.
Phase 2: Between-group differences of age distribution | At enrollment.
  Data on age will be presented as mean ± standard deviation and the independent t-test will be applied to investigate between-group differences (single patients vs. patients in a relationship vs. partner/spouse).
Phase 2: Between-group differences in gender distribution | At enrollment.
  Data on sex will be presented as frequency with percentage using. Chi Square test will be applied to investigate between-group differences (single patients vs. patients in a relationship vs. partner/spouse).
Phase 2: Between-group differences in educational level | At enrollment.
  Data on educational level will be presented as frequency with percentages. Chi Square test will be applied to investigate between-group differences (single patients vs. patients in a relationship vs. partner/spouse).
Phase 2: Between-group differences in disease stage | At enrollment.
  Data on disease stage by Leibovich disease risk groups (low, medium, and high) be presented as frequency and percentages. To investigate between-group differences (single patients vs. patients in a relationship) the Chi Square test will be applied
Phase 2: Between-group differences of comorbidity burden | At enrollment.
  The Charlson Comorbidity Index will be applied to investigate disease burden in single patients versus non-single patients. The higher the score, the worse the prognosis.
  0 points: No comorbidities are present. 1-2 points: Moderate comorbidity. 3 points or above: Severe comorbidity. Data will be presented as frequency and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta R Villumsen, PhD, Study Chair — Gødstrup Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Gødstrup Hospital, Herning

IPD SHARING:
Plan to Share IPD: Undecided
Yet to be discussed in the steering group

REFERENCES:
- [Background] Hamilton CB, Hoens AM, McKinnon AM, McQuitty S, English K, Hawke LD, Li LC. Shortening and validation of the Patient Engagement In Research Scale (PEIRS) for measuring meaningful patient and family caregiver engagement. Health Expect. 2021 Jun;24(3):863-879. doi: 10.1111/hex.13227. Epub 2021 Mar 17. PMID 33729634
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Roberts JP, Fisher TR, Trowbridge MJ, Bent C. A design thinking framework for healthcare management and innovation. Healthc (Amst). 2016 Mar;4(1):11-4. doi: 10.1016/j.hjdsi.2015.12.002. Epub 2016 Jan 14. PMID 27001093
- [Background] Altman M, Huang TTK, Breland JY. Design Thinking in Health Care. Prev Chronic Dis. 2018 Sep 27;15:E117. doi: 10.5888/pcd15.180128. PMID 30264690
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Smith A', Wu VS, Lambert S, Lamarche J, Lebel S, Leske S, Girgis A. A systematic mixed studies review of fear of cancer recurrence in families and caregivers of adults diagnosed with cancer. J Cancer Surviv. 2022 Dec;16(6):1184-1219. doi: 10.1007/s11764-021-01109-4. Epub 2021 Nov 11. PMID 34762248
- [Background] Bergerot CD, Battle D, Philip EJ, Bergerot PG, Msaouel P, Smith A', Bamgboje AE, Shuch B, Derweesh IH, Jonasch E, Stern AP, Pal SK, Staehler M. Fear of Cancer Recurrence in Patients With Localized Renal Cell Carcinoma. JCO Oncol Pract. 2020 Nov;16(11):e1264-e1271. doi: 10.1200/OP.20.00105. Epub 2020 Sep 18. PMID 32955409